CLINICAL TRIAL: NCT01951339
Title: Impact of Sitagliptin on Cardiovascular Exercise Performance in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 13-2015
Record Dates: First submitted 2013-09-19; First posted 2013-09-26 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes; Cardiovascular Disease
Keywords: diabetes; type 2 diabetes; exercise; echo; heart; sitagliptin; glimepiride; cardiovascular
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus; Motor Activity | interventions — Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | US Export: Yes

ARMS (2):
- Sitagliptin plus placebo (Experimental): 100 mg sitagliptin plus 2 mg placebo once daily for three months
  Interventions: Drug: Sitagliptin; Drug: Placebo
- Glimepiride plus placebo (Active Comparator): 2 mg glimepiride plus 100 mg placebo once daily for three months
  Interventions: Drug: Glimepiride; Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — 100 mg sitagliptin
  Other Names: Januvia (sitagliptin)
  Arms: Sitagliptin plus placebo
Drug: Glimepiride — Active Comparator
  2mg glimepiride
  Other Names: Amaryl
  Arms: Glimepiride plus placebo
Drug: Placebo — 2 mg placebo once daily
  Other Names: Placebo 1-sitagliptin
  Arms: Sitagliptin plus placebo
Drug: Placebo — 100 mg placebo once daily for three months
  Other Names: Placebo 2- glimepiride
  Arms: Glimepiride plus placebo

SUMMARY:
The goal of this study is to examine whether sitagliptin, an agent which enhances the action of hormones that control the release of insulin and is already in clinical use for type 2 diabetes, might also improve functional exercise capacity.

Specific aims:

1. To test whether sitagliptin will improve functional exercise capacity in persons with type 2 diabetes compared to glimepiride.

1a. The primary outcome will be peak oxygen consumption (VO2peak) and oxygen uptake kinetics (VO2 kinetics).

1b. Secondary outcomes include cardiac function, endothelial function and tissue oxygen saturation (STO2) as well as health-related quality of life.

2. To evaluate the impact of sitagliptin on muscle mitochondrial function 2a. The primary outcome to address this aim will be 31P measurements (phosphocreatine, free inorganic phosphate, adenosine triphosphate peaks, adenosine diphosphate and pH)

Impact: Novel approaches are needed to decrease excess cardiovascular morbidity and mortality in diabetes. Diabetes impairs cardiovascular fitness and thereby mortality. A demonstration that sitagliptin improves cardiovascular fitness, (and possibly mitochondrial function) will provide important new data pertinent to the management of diabetes and pre-diabetes.

DETAILED DESCRIPTION:
Subjects will come for a total of nine testing visits during which evaluations will take place. Visits are structured as follows:

1. After subjects review the study and give consent for study participation, a history and physical exam will be performed. Ankle brachial index, autonomic nervous system function tests, the Low-level Physical Activity Recall questionnaire and vital signs will be performed.
2. Blood drawn for measurement of hemoglobin A1C, fasting glucose, fasting insulin, free fatty acids and microalbuminuria, c-reactive protein, interleukin 6, adiponectin, and creatinine and glycerol. Additional screening labs include complete blood count (CBC), follicle-stimulating hormone, urine protein and a lipid panel to assess whether women are pre- or post-menopausal (FSH), and overall health (CBC, lipids and urine protein). A dietary survey will be administered for food preferences for the three day study diet administered prior to visits 3-5 and 7-9. Dual-energy xray absorptiometry (DEXA) and body composition tests will be done to ensure that groups are weight similar (using fat-free mass). A pulmonary function test, resting electrocardiogram (EKG) and familiarization bicycle test will be performed.
3. Subjects will receive a three day study diet prior to visit 3. A resting and exercise EKG will be performed on the day of the visit. A graded exercise test will be done to determine the VO2peak. Patients will have measures of cardiac function and endothelial function on visit 3 by plethysmography and cardiac echo. Vital signs will be taken at rest.
4. Subjects will receive a three day study diet prior to visit 4. Calf muscle magnetic resonance spectroscopy (MRS) will be performed on a 3.0 T whole-body MRI scanner.
5. During visit 5, arterial stiffness/endothelial function will be non-invasively measured by the Sphygmocor system. Subjects will also have three constant-load tests to measure VO2 kinetics where oxygen saturation (StO2) will be measured during exercise. A resting and exercise EKG and vital signs will be performed during the visit. Subjects will be randomized to taking sitagliptin plus placebo or glimepiride plus placebo and all must be taking metformin (1-2 grams /d) for 3 months. Sitagliptin and its placebo will be administered 100 mg/d. Glimepiride and its placebo will be administered 2 mg/day. During the treatment phase subjects will be given a log to keep track of their blood glucose each day.
6. Visit 6 will consist of a physical exam with a clinician as well as a blood draw and check of vital signs during sitagliptin or glimepiride treatment.
7. After 3 months of sitagliptin or glimepiride administration, Visit 3 will be repeated. Additional testing to be performed during visit 7 will include a physical exam performed by a study physician, blood work for covariate lab tests listed in Visit 2 and the Low-level Physical Activity Recall(LoPAR) questionnaire.
8. During visit 8, visit 4 procedures will be repeated.
9. During visit 9, the testing performed during visit 5 will be repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects may be pre, peri or post-menopausal.
2. People who do not participate in a regular exercise program (> one bout of exercise per week).
3. Presence of type 2 diabetes will be documented by chart review that will confirm the diagnosis as well as the presence of treatment for diabetes.
4. Persons with type 2 diabetes will be accepted for study only if they have total glycosylated hemoglobin levels (HbA1C) between 7 and 9.5% (adequate control) on therapy.
5. Persons who are taking metformin 500-2000 mg/day only to control their T2D, but are not taking any other diabetes medication in addition to or instead of metformin.
6. Persons not taking medication to control diabetes.

Exclusion Criteria:

1. Females of childbearing potential who are pregnant, planning to become pregnant or breastfeeding.
2. Persons will be excluded if they have evidence of ischemic heart disease by history or abnormal resting or exercise electrocardiogram (EKG) (> 1 mm ST segment depression), regional wall motion abnormalities, left ventricular systolic dysfunction or significant valvular disease.
3. Persons with angina or any other cardiac or pulmonary symptoms potentially limiting exercise performance.
4. Presence of systolic blood pressure >190 at rest or >250 with exercise or diastolic pressure >95 at rest or >115 with exercise.
5. Subjects who have peripheral arterial disease.
6. Subjects with proteinuria (urine protein >200 mg/dl) or a creatinine > 2 mg/dl, suggestive of renal disease.
7. Persons with liver function impairment defined as elevated liver function tests three times the upper limit.
8. Persons with a history of pancreatitis.
9. Subjects more than 140% of ideal body weight.
10. Patients on insulin therapy will not be included.
11. Current smokers will not be accepted for study since smoking can impair cardiovascular exercise performance but people who have quit smoking for at least 1year will be accepted for study.
12. Persons with autonomic dysfunction (>20 mm fall in upright blood pressure without a change in heart rate) will be excluded.
13. Diabetic persons with clinically evident distal symmetrical neuropathy will be excluded from further study, because of possible effects on exercise performance, by evaluation of symptoms (numbness, paresthesia) and signs (elicited by vibration, pinprick, light touch, ankle jerks).
14. Persons with diabetic ketoacidosis.
15. Persons with a serious hypersensitivity to sitagliptin, sulfonylureas or sulfonamides.
16. Inability to walk or ride a bike unassisted for a continuous 5 minutes.
17. Subjects will be excluded if they have any implanted metal in their body.
18. Subjects currently being treated with Digoxin.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith G. Regensteiner, PhD, Principal Investigator — University of Colorado, Denver; Jane EB Reusch, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scalzo RL, Rafferty D, Schauer I, Huebschmann AG, Cree-Green M, Reusch JEB, Regensteiner JG. Sitagliptin improves diastolic cardiac function but not cardiorespiratory fitness in adults with type 2 diabetes. J Diabetes Complications. 2019 Aug;33(8):561-566. doi: 10.1016/j.jdiacomp.2019.05.002. Epub 2019 May 10. PMID 31182338

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients underwent screening, as well as baseline data collection prior to randomization to group. Several patients withdrew from the study prior to randomization.
Groups:
- Glimepiride Plus Placebo: 2 mg glimepiride plus 100 mg placebo once daily for three months
  Glimepiride: Active Comparator
  2mg glimepiride
  Placebo: 100 mg placebo once daily for three months
Period: Overall Study
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Started | 15 | 15
Completed | 13 | 14
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (2) | 57 (3) | 57 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 1 | 5
  White | 8 | 13 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Peak Oxygen Consumption (VO2peak).
Description: Subjects' peak oxygen consumption will be tested on a stationary bike before and after 3 months of study medication.
Time Frame: Pre-intervention (Baseline) and post-intervention (3 months)
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Number analyzed (Participants) | 13 | 14
ml/min
  Pre-intervention | 1893 (138) | 1953 (113)
  Post-intervention | 1849 (135) | 1881 (151)

2. Primary Outcome: Changes From Baseline in 31P Measurement: Phosphocreatine Time Constant
Description: Potential change in muscle mitochondrial function will be assessed after three months of study medication treatment
Time Frame: Pre-intervention (Baseline) and post-intervention (3 months)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Number analyzed (Participants) | 7 | 8
seconds
  Pre-intervention | 34.1 (7.3) | 30.9 (3.9)
  Post-intervention | 26.6 (2.9) | 29.6 (3.6)

3. Primary Outcome: Change in Oxygen Uptake Kinetics (VO2 Kinetics)
Description: Oxygen uptake kinetics will be tested on a stationary bike before and after 3 months of study medication. VO2 kinetics is reported as the time constant associated with the change in oxygen update from rest to steady state.
Time Frame: Pre-intervention (Baseline) and post-intervention (3 months)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Number analyzed (Participants) | 13 | 14
seconds
  Pre-intervention | 56.2 (5.0) | 54.2 (7.3)
  Post-intervention | 67.5 (8.0) | 54.6 (4.3)

4. Primary Outcome: Changes From Baseline in 31P Measurement: Free Pi Time Constant
Description: Potential change in muscle mitochondrial function will be assessed after three months of study medication treatment. Data are represented as the change in Pi through the scan.
Time Frame: Pre-intervention (Baseline) and post-intervention (3 months)
Population: These data are quality control measures only.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Number analyzed (Participants) | 14 | 15
seconds
  Pre-intervention | 29.73 (10.16) | 28.54 (10.44)
  Post-intervention | 27.94 (3.82) | 26.15 (5.60)

5. Primary Outcome: Changes From Baseline in 31P Measurement: Adenosine Triphosphate (ATP) Peaks
Description: Potential change in muscle mitochondrial function will be assessed after three months of study medication treatment
Time Frame: Pre-intervention (Baseline) and post-intervention (3 months)
Population: These data are quality control measures only.
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Number analyzed (Participants) | 14 | 15
mM
  Pre-intervention | 8.19 (0.22) | 7.93 (0.58)
  Post-intervention | 12.66 (13.59) | 8.02 (0.29)

6. Primary Outcome: Changes From Baseline in 31P Measurement: Adenosine Diphosphate (ADP) Time Constant
Description: Potential change in muscle mitochondrial function will be assessed after three months of study medication treatment
Time Frame: Pre-intervention (Baseline) and post-intervention (3 months)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Number analyzed (Participants) | 7 | 8
seconds
  Pre-intervention | 28.0 (5.3) | 24.5 (3.5)
  Post-intervention | 19.4 (1.1) | 21.2 (2.9)

7. Primary Outcome: Changes From Baseline in 31P Measurement: pH
Description: Potential change in muscle mitochondrial function will be assessed after three months of study medication treatment
Time Frame: Pre-intervention (Baseline) and post-intervention (3 months)
Population: These data are quality control measures only.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Number analyzed (Participants) | 14 | 15
pH
  Pre-intervention | 6.88 (0.05) | 6.88 (0.05)
  Post-intervention | 6.85 (0.02) | 6.89 (0.05)

8. Secondary Outcome: Changes From Baseline in Echocardiographic Measures (Stroke Volume)
Description: Potential change in cardiac function will be assessed by echocardiography before and after 3 months of study medication
Time Frame: Pre-intervention (Baseline) and post-intervention (3 months)
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Number analyzed (Participants) | 13 | 14
mL/beat
  Pre-intervention | 58.2 (5.5) | 72.7 (6.1)
  Post-intervention | 64.6 (11.9) | 77.8 (6.7)

9. Secondary Outcome: Change in (Non-invasively Measured) Deoxygenated Hemoglobin Concentration in the Vastus Lateralis During Exercise
Description: Deoxygenated hemoglobin concentration will be measured using near-infrared spectroscopy during sub-maximal exercise before and after 3 months of study drug administration.
Time Frame: Pre-intervention (Baseline) and post-intervention (3 months)
Population: This variable was listed as a secondary outcome of the study that was later dropped by the investigators after a careful review of the literature. We decided not to pursue this outcome because it was not scientifically useful to address the original hypothesis.
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during individual study participation, approximately 6 months.
Arm/Group | Sitagliptin Plus Placebo | Glimepiride Plus Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin Plus Placebo (N=15) | Glimepiride Plus Placebo (N=15)
Medication side effects (Gastrointestinal disorders) | 3 (3) | 1 (1)
High blood glucose (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Mild hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT01951339/Prot_SAP_000.pdf